CLINICAL TRIAL: NCT05228795
Title: Value of Glypican-1 Expression in Pleural Epithelioid Mesothelioma, Adenocarcinoma and Squamous Cell Carcinoma of the Lung
Brief Title: Glypican-1 Expression in Epithelioid Mesothelioma, Adenocarcinoma and SCC of the Lung
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nagwa Abd El-Sadek Ahmed, Lecturer at Pathology Department, Faculty of Medicine, Sohag University, Sohag University
Other Study IDs: Soh-Med-22-01-29
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer Adenocarcinoma; Lung Cancer Squamous Cell; Mesothelioma; Lung
Keywords: Glypican-1; Epitheloid mesothelioma; Lung adenocarcinoma; Lung SCC
MeSH Terms: conditions — Adenocarcinoma of Lung; Mesothelioma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung carcinoma is the second most common cancer and a leading cause of cancer-related mortality worldwide. In Egypt, lung carcinoma ranks the 5th among all cancer cases. Malignant mesothelioma is an aggressive neoplasm that arises from mesothelial cells which form the lining of the pleural. There is a strong resemblance between epithelioid mesothelioma and lung adenocarcinoma, some of peripheral lung adenocarcinoma or SCC present with pleurotropic growth like mesothelioma. Glypican-1 (GPC1) is one the six glypican family members. It is one of cell surface heparan sulfate proteoglycans that acts as a growth factor signaling. The aim of this study is to evaluate the immunohistochemical expression of Glypican-1 in pleural epitheloid mesothelioma, lung adenocarcinoma and lung SCC

DETAILED DESCRIPTION:
Lung carcinoma is the second most common cancer and a leading cause of cancer-related mortality worldwide, comprising almost 20% of all cancer deaths. In Egypt, lung carcinoma ranks the 5th among all cancer cases. It is more common in males than females, and most people diagnosed at the age of 65 years or older. The main risk factor of lung malignancy is tobacco smoking.

There are two main histologic variants of lung carcinoma, non-small cell lung cancer (NSCLC) and small-cell lung cancer (SCLC). NSCLC represents more than 80% of all lung carcinomas. Histologically, NSCLC is divided into adenocarcinoma, squamous cell carcinoma (SCC) and large cell carcinoma; of which lung adenocarcinoma is the most common subtype representing about 40%. Specific therapies can be offered to patients based on the histological and molecular status of primary tumors. Therefore, an accurate differentiation between solid predominant lung adenocarcinoma and poorly differentiated lung SCC has become increasingly indispensable; the accurate discrimination of these two main histological types is required for gene-targeted therapy.

Malignant mesothelioma is an aggressive neoplasm that arises from mesothelial cells which form the lining of the pleural, pericardial, and peritoneal cavities. Majority of malignant mesothelioma, approximately 85%, occur in pleural cavity and most of the remainder arising in the peritoneum. In the United States around 3,000 new cases are diagnosed each year. In Egypt, pleural malignant tumors formed 1.3% of total malignant tumors. Pleural mesothelioma is the most frequent primary pleural malignant tumor forming more than half of the cases. The main risk factor for pleural mesothelioma is exposure to asbestos. Other risk factors may include; radiation exposure, old age, male gender and exposure to certain other minerals.

Malignant mesothelioma is divided into three histologic variants that include: epithelioid, sarcomatoid and biphasic variants. Epithelioid variant is the most common subtype representing 70% of malignant mesothelioma. There is a strong resemblance between epithelioid mesothelioma and lung adenocarcinoma, some of peripheral lung adenocarcinoma or SCC present with pleurotropic growth like mesothelioma. The prognosis and management of epithelioid mesothelioma differ from lung carcinoma, so accurate diagnosis of mesothelioma is necessary.

Glypican-1 (GPC1) is one the six glypican family members. It is one of cell surface heparan sulfate proteoglycans that acts as a growth factor signaling. It plays role in the control of cell division and growth regulation. It is encoded by GPC1 gene located at 2q37. It contains 588 amino acids with three predicted heparan sulfate chains. It has been evaluated as a potential target for cancer therapy. Many studies have shown that GPC1 is crucial for efficient cancer cell growth, metastasis and angiogenesis. Glypican-1 overexpression has previously been reported in breast cancer, pancreatic cancer and glioma.

Studies evaluating the expression of Glypican-1 in pleural mesothelioma and lung carcinoma are deficient. Knowledge about its potential value in differentiation between pleural epithelioid mesothelioma, lung adenocarcinoma and SCC needs further elucidation.

Aim of This Work:

The aim of this study is to evaluate the immunohistochemical expression of Glypican-1 in pleural epitheloid mesothelioma, lung adenocarcinoma and lung SCC, and to correlate its expression with some known clinico-pathological parameters, to evaluate its diagnostic and prognostic role.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pleural epithelioid mesothelioma and lung adenocarcinoma and SCC who underwent surgery

Exclusion Criteria:

* Patients received pre-operative chemotherapy or radiotherapy.
* Patients with insufficient clinical data.
* Specimens with extensive necrosis
* Tiny specimens which are insufficient for accurate diagnosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: sixty specimens including: 20 cases of pleural epitheloid mesothelioma, 20 cases of lung adenocarcinoma and 20 cases of lung SCC obtained from patients who underwent excisional biopsy in Cardiothoracic Department, according to local Ethical Committee regulations, to be examined in the Pathology Laboratory of Sohag Faculty of Medicine. From January 2022 till completing the sample size.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
evaluate the immunohistochemical expression of Glypican-1 in pleural epitheloid mesothelioma, lung adenocarcinoma and lung SCC | 1 month
  Immunohistochemical study
to correlate its expression with some known clinico-pathological parameters, to evaluate its diagnostic and prognostic role. | 1 month
  Statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Ahmed, Lecturer, Principal Investigator — Sohag University
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt